CLINICAL TRIAL: NCT02168257
Title: Neotech RAM Cannula Versus Conventional Binasal Prong Continuous Positive Airway Pressure (CPAP) to Treat Respiratory Distress in Low Birth Weight Neonates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1303-032; 47575 (Other Grant/Funding Number: Children's Hospitals and Clinics of Minnesota IRGP)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Distress Syndrome, Newborn; Continuous Positive Airway Pressure; Low Birth Weight Infants
Keywords: Nasal Cannula
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAM Cannula CPAP (Experimental): CPAP provided by RAM Cannula
  Interventions: Device: RAM Cannula
- Binasal Prong CPAP (Active Comparator): CPAP provided by binasal prong
  Interventions: Device: Binasal Prong CPAP

INTERVENTIONS:
Device: RAM Cannula
  Arms: RAM Cannula CPAP
Device: Binasal Prong CPAP
  Arms: Binasal Prong CPAP

SUMMARY:
The purpose of this study is to determine if the RAM cannula is as effective as conventional binasal prongs to deliver CPAP to low birth weight infants with respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Low Birth Weight Infant
* Currently on continuous positive aireway pressure of 5-7 cm water pressure
* Receiving continuous positive airway pressure support for > 24 hrs prior to enrollment
* Fraction of inspired oxygen requirement of 23-50%

Exclusion Criteria:

* Fraction of inspired oxygen > 50%
* Congenital defects of head, pulmonary or cardiovascular systems
* Chromosomal abnormalities/genetic syndromes
* Invasive Surgical Procedure within 24 hrs prior to enrollment
* Enrollment in separate clinical trial that has ongoing data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Oxygenation | 3 hrs
  Pulse oximetry
Ventilation | 3 hrs
  transcutaneous carbon dioxide monitor

SECONDARY OUTCOMES:
Esophageal pressure measurements | 3 hrs
  Esophageal Pressure Catheter
Apnea | 3 hrs
  3-channel pneumogram

OTHER OUTCOMES:
Pulse | 3 hrs
Respiratory Rate | 3 hrs
Blood Pressure | 3 hrs
Oxygen requirement | 3 hrs
  Measured by fraction of inspired oxygen to maintain target pulse oximetry saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Neil P Mulrooney, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota; Andrea L Lampland, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota, United States